CLINICAL TRIAL: NCT05618535
Title: Effect of Body Position on Hemodynamics in Patients With Acute Ischemic Stroke Undergoing Ultra-early Reperfusion Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of The First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EBPHPAIS-URT
Record Dates: First submitted 2022-11-10; First posted 2022-11-16 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zero position (Sham Comparator): All monitoring was done from 9 to 11 a.m., and the whole monitoring process was carried out in a specific and quiet environment at 20-24℃ to avoid other auditory and visual stimuli. After 10min of the relaxed supine position, the blood pressure, heart rate, and blood flow velocity of the middle cerebral artery were measured in the 0° position for 5min.
  Interventions: Device: Transcranial Doppler.
- 30 degrees position (Experimental): Within 30 seconds after the 0° position measurement completion, the subjects were transferred to the 30° position and rested for 15 minutes under the 30° position. In other words, a washout period of 15 minutes was established between two measurements to ensure the stability of vital signs and avoid confounding effects. The blood pressure, heart rate, and blood flow velocity of the middle cerebral artery were measured again for 5 minutes after the vital signs were stable.
  Interventions: Device: Transcranial Doppler.

INTERVENTIONS:
Device: Transcranial Doppler. — Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size.
  Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler.

SUMMARY:
The aim of this study was to determine the differences in hemodynamics between different positions in patients undergoing ultra-early reperfusion therapy.

DETAILED DESCRIPTION:
Hemodynamic stability can prevent hypoperfusion or hyperperfusion after reperfusion therapy. It has been reported in a large number of literatures that body position has an effect on hemodynamics, but the effect of different body positions on the hemodynamics of patients undergoing ultra-early reperfusion therapy is not clear. In this study, we hypothesized that the hemodynamics of patients undergoing ultra-early reperfusion therapy would differ between different positions.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years, < 80 years, regardless of sex；
* Patients with clinically confirmed acute ischemic stroke who received intravenous thrombolysis or emergency endovascular treatment;
* Baseline National Institute of Health stroke scale（NIHSS）score ≤25;
* Baseline Glasgow Coma Scale (GCS) ≥8;
* Signed and dated informed consent is obtained

Exclusion Criteria:

* The patient has clear indications or contraindications, such as active vomiting, spinal cord injury；
* Clinicians considered that the assigned body position could not be maintained; Patients unable to cooperate with all noninvasive beat-by-beat continuous BP monitoring;
* Poor temporal window penetration;
* Patients with diseases that seriously affect hemodynamics, such as atrial fibrillation, anemia, and hyperthyroidism;
* Previous history of atrial fibrillation or ECG showing atrial fibrillation or arrhythmia;
* Pregnant or lactating women;
* Poor treatment compliance;
* Complicated with severe systemic diseases, such as heart failure, respiratory failure, renal failure, gastrointestinal bleeding, coagulopathy, malignant tumors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Differences in blood pressure variability（BPV）between different positions | 0-7 days
  BPV is defined as blood pressure oscillations in relation to the mean values.
Differences in heart rate variability (HRV) between different positions | 0-7 days
  HRV is defined as heart rate oscillations in relation to the mean values.

SECONDARY OUTCOMES:
The difference of middle cerebral artery blood flow velocity between different positions. | 0-7 days
  Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China